CLINICAL TRIAL: NCT06898606
Title: Psilocybe Cubensis Mushrooms With or Without Fluoxetine for Refractory Depression: a Phase 2a Pilot Randomized Clinical Trial (COGUNILA)
Acronym: COGUNILA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Federal University of Latin American Integration (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COGUNILA; CAAE: 77979424.0.0000.0107 (Registry Identifier: BRAZIL PLATFORM)
Record Dates: First submitted 2024-11-30; First posted 2025-03-27 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Depressive Disorder
Keywords: Psilocybin; Depression; Fluoxetine; Treatment; Psychedelics
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — Psilocybin; Fluoxetine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel-group trial in adults with treatment-resistant major depressive disorder. All participants receive one psychedelic-assisted session with 3g of Psilocybin musshoroms and psychotherapy; they are randomized to concurrent daily fluoxetine 20 mg or matching placebo for 4 weeks (started 2 weeks before dosing and continued 2 weeks after). The study compares psychedelic experience, antidepressant effects, and adverse events between arms.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psilocybin + Fluoxetine (Experimental): 2 preparation sessions for the psychedelic experience
  1. dosing session with 3g Psilocybe mushrooms (single oral dose), with psychotherapy assistance
  2. integration sessions Fluoxetine 20 mg/day for 4 weeks (started 2 weeks before dosing and continued 2 weeks after)
  Interventions: Drug: Psilocybin and Psilocyn; Behavioral: Psychotherapy-assisted session; Drug: Fluoxetine
- Psilocybin + Placebo (Placebo Comparator): 2 preparation sessions for the psychedelic experience
  1. dosing session with 3g Psilocybe mushrooms (single oral dose), with psychotherapy assistance
  2. integration sessions Pharmaceutical grade talc, matching placebo (identical capsules), daily for 4 weeks (started 2 weeks before dosing and continued 2 weeks after).
  Interventions: Drug: Psilocybin and Psilocyn; Drug: Placebo; Behavioral: Psychotherapy-assisted session

INTERVENTIONS:
Drug: Psilocybin and Psilocyn — Oral dose administered via Psilocybe mushrooms material batch-assayed by LC-MS to standardize psilocybin and psilocyn content.
Drug: Placebo — Matching capsules, once daily for 4 weeks (-14 to +14 days).
  Arms: Psilocybin + Placebo
Behavioral: Psychotherapy-assisted session — Same manualized procedures as Arm 1.
Drug: Fluoxetine — 20 mg/day for 4 weeks (-14 to +14 days relative to dosing day).
  Arms: Psilocybin + Fluoxetine

SUMMARY:
This Phase 2a pilot, exploratory, randomized, double-blind, placebo-controlled, parallel-group trial will estimate whether concurrent fluoxetine alters the antidepressant effect, acute psychedelic experience, or safety of a psychedelic-assisted psychotherapy session in adults with treatment-resistant major depressive disorder (TRD). Eligible participants (ages 25-64) have DSM-5-TR MDD, moderate-severe, MADRS ≥20, and partial response in the current episode (≥1 adequate antidepressant trial of 6-12 weeks with <50% symptom reduction). All participants receive one dosing session with 3g of standardized Psilocybe mushrooms - with batch assay (e.g., LC-MS) to determine the amount of psilocybin and psilocin present in the sample - with manualized preparation and integration. Participants are randomized 1:1 to fluoxetine 20 mg/day or matching placebo for 4 weeks, started 2 weeks before the psychedelic session and continued 2 weeks after. Masking is quadruple (participant, care provider, investigator, outcomes assessor). The primary outcome is change in MADRS from Baseline to Week 4, assessed by a remote, blinded rater. Key secondary outcomes include response (≥50% MADRS reduction) and remission (MADRS ≤10) at Week 4, and durability at Week 6. Exploratory outcomes assess the psychedelic experience (5D-ASC, SOCQ), psychological flexibility (AAQ-10), and safety/tolerability (UKU and adverse events). Findings will be interpreted as estimates with 95% confidence intervals to inform the design of a subsequent confirmatory trial.

DETAILED DESCRIPTION:
This is a Phase 2a pilot, exploratory, randomized, double-blind, placebo-controlled, parallel-group clinical trial designed to estimate the effect of concurrent fluoxetine on the efficacy, acute psychedelic experience, and safety of a psychedelic-assisted psychotherapy session in adults with treatment-resistant major depressive disorder (TRD).

Rationale. Selective serotonin reuptake inhibitors (SSRIs) rapidly increase synaptic 5-HT via SERT blockade (days), whereas receptor-level adaptations (e.g., 5-HT2A down-regulation/desensitization) typically require weeks. By administering the psychedelic session after 2 weeks of fluoxetine (and continuing fluoxetine for 2 additional weeks), the study primarily probes the impact of SERT blockade per se on the psychedelic experience and antidepressant outcomes, while minimizing later, slower receptor adaptations. The design-psychedelic for both arms with blinding of fluoxetine vs matching placebo-also improves masking compared with classic "psychedelic vs placebo" trials and directly addresses the practical question of whether SSRI co-administration attenuates, has no meaningful impact, or improves tolerability.

Participants and eligibility. Adults ≥25 and <65 years with current DSM-5-TR MDD, moderate to severe, confirmed by SCID-5, and MADRS ≥20 at baseline. TRD is defined here as Partial Response in the current episode: ≥1 adequate antidepressant trial (therapeutic dose for ≥6-12 weeks, adherence ≥80%) with <50% symptom reduction or clinically significant residual symptoms. Key exclusions include bipolar/psychotic disorders (personal) or first-degree family history, acute suicide risk, contraindications to study medications, unstable medical illness, and current use of serotonergic agents that cannot meet protocol-defined washout. (Full Inclusion/Exclusion lists appear in the Eligibility section.)

Interventions. All participants receive a single psychedelic-assisted session with manualized preparation (2 sessions), dosing-day support, and integration (2 sessions). Administration will be carried out with 3g of standardized Psilocybe mushrooms for all participants, with batch assay (e.g., LC-MS) to determine the amount of psilocybin and psilocin present in the sample. Participants are randomized 1:1 to:

Fluoxetine 20 mg/day for 4 weeks (started 2 weeks before the psychedelic session and continued 2 weeks after), or Matching placebo for 4 weeks on the same schedule. Randomization and masking. Allocation is randomized 1:1, stratified by baseline severity (MADRS 20-29 vs ≥30) using permuted blocks of variable size. Masking is quadruple (participants, care providers, investigators, and outcome assessors). Fluoxetine and placebo are provided in identical capsules; blinding integrity is assessed post-dose and at Week 4 (guess + confidence).

Assessments and instruments. Depressive symptoms are measured primarily with MADRS (Baseline, Week 1, Pre-dose/Week 2, Week 4, Week 6). For characterization/triage, HAM-D-21 may be used at baseline. The psychedelic experience is measured with 5D-ASC (6-24 h post-dose) and SOCQ (~24 h post-dose). Psychological flexibility is assessed with AAQ-10 (Baseline, Week 4, Week 6). Safety is captured with the UKU Side Effect Rating Scale at Baseline, Week 1, Pre-dose/Week 2, 24-48 h post-dose, Week 4, Week 5 and Week 6; adverse events and serious adverse events are recorded throughout.

Outcome measures. Primary outcome: Change in MADRS total score from Baseline to Week 4. Key secondary outcomes: Response (≥50% MADRS reduction) at Week 4; Remission (MADRS ≤10) at Week 4; durability (Baseline→Week 6 change); UKU totals/subscales and incidence of adverse events (any, moderate-severe) and serious adverse events.

Exploratory outcomes: 5D-ASC total/domains and proportion meeting "complete mystical experience"; SOCQ selected domains; AAQ-10 changes (Baseline→Week 4/6); correlations between psychedelic-experience metrics and antidepressant outcomes; comparative profiles of adverse effects between arms.

Statistical approach. The primary analysis compares arms using ANCOVA for Week-4 MADRS, adjusting for baseline MADRS (continuous). Results are presented as adjusted mean difference, 95% confidence interval, and standardized effect size (e.g., Hedges g). Given the pilot nature (N=24), inference is estimative rather than confirmatory; findings are interpreted with reference to a clinically meaningful margin for exploratory non-inferiority (e.g., -4 MADRS points). Secondary and exploratory outcomes are summarized with effect estimates and 95% CIs; p-values, if reported, are descriptive. A linear mixed model using all time points may be used as a sensitivity analysis for missing data assumed missing-at-random.

Safety and oversight. Safety monitoring includes systematic UKU assessments and continuous adverse-event surveillance from consent through Week 6, with prespecified criteria for temporary interruption or discontinuation. Concomitant medications that could compromise masking or interact serotonergically are restricted per protocol; permitted rescue options and timing windows are specified to protect outcome integrity.

This Phase 2a pilot aims to inform feasibility, mechanism, and effect size by directly testing whether concurrent fluoxetine meaningfully alters the acute psychedelic experience, antidepressant response, or tolerability/safety of psychedelic-assisted therapy in TRD.

ELIGIBILITY:
Inclusion Criteria Age: ≥25 and <65 years. Diagnosis: Current Major Depressive Disorder (MDD), moderate to severe, per DSM-5-TR, confirmed with SCID-5.

Baseline severity: MADRS ≥20 at baseline (reassessed at the pre-dose visit to confirm ongoing eligibility).

Partial Response in the current episode (PRD): ≥1 adequate antidepressant trial in this episode (therapeutic dose for ≥6-12 weeks, adherence ≥80%) with <50% symptom reduction or clinically significant residual symptoms.

Clinical stability and ability to provide informed consent; willingness to comply with all study procedures (preparation, dosing session, integration, and follow-ups).

Contraception: For participants with reproductive potential, negative pregnancy test and agreement to use effective contraception during the study.

Exclusion Criteria Psychiatric disorders: Bipolar I/II disorder, any psychotic disorder, or current MDD with psychotic features; first-degree family history of psychotic or bipolar disorder.

Suicide risk: Acute suicidal risk, e.g., active suicidal ideation with intent or plan, recent attempt, or clinical judgment requiring urgent intervention.

Interacting medications: Current use of serotonergic antidepressants (SSRI/SNRI/MAOI, clomipramine) or other pro-serotonergic agents (e.g., triptans, linezolid, lithium, tramadol, dextromethorphan) that cannot be discontinued per protocol-defined washout.

Other psychotropics: Unstable doses of antipsychotics, mood stabilizers, or long-acting benzodiazepines within the last 2 weeks; need for medications that would compromise blinding on the dosing day.

Psychotherapy changes: Initiation or major change in psychotherapy within 2 weeks prior to baseline (to preserve clinical stability).

Medical conditions: Clinically significant or unstable medical illness (cardiovascular, neurological, hepatic, renal), prolonged QTc, known hypersensitivity/contraindication to fluoxetine or study materials.

Pregnancy or breastfeeding. Substance use: Current substance use disorder (excluding nicotine/caffeine) within the past 3 months; non-medical cannabis use that cannot meet the pre-dose abstinence window (e.g., ≥72 h).

Any condition that, in the investigator's opinion, would make participation unsafe or interfere with the assessments.

Washout note (to include in Procedures/Eligibility):

SSRIs/SNRIs: 7 days or ≥5 half-lives; prior fluoxetine: ≥6 weeks; MAOIs: ≥14 days before randomization/dosing. Participants must be willing and able to follow the washout schedule.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
Change in MADRS Total Score | 4 weeks
  The primary antidepressant outcome is the change in Montgomery-Åsberg Depression Rating Scale (MADRS) total score from baseline (Day 0) to Week 4. MADRS ranges 0-60 (higher = more severe). Interviews will be conducted by a remote, blinded, independent assessor using the structured interview guide at Baseline, Week 1, Pre-dose (Week 2), Week 4 and Week 6. The primary contrast will be the adjusted difference between arms at Week 4 (ANCOVA controlling for baseline MADRS); effect size and 95% CI will be reported.

SECONDARY OUTCOMES:
MADRS Response | 4 week
  Proportion of participants achieving ≥50% reduction in MADRS total score from baseline to Week 4.
MADRS Remission | 4 week
  Proportion of participants with MADRS total score ≤10 at Week 4.
Durability of Antidepressant Effect | 6 week
  Change in MADRS total score from baseline to Week 6.
Adverse Effects - UKU | Baseline; Week 1; Pre-dose (Week 2); 24-48 h post-dose; Week 4; Week 6
  UKU Side Effect Rating Scale total and subscales (psychic, neurologic, autonomic, sexual); incidence of adverse events (any; moderate-severe) and serious adverse events.

OTHER OUTCOMES:
Quality of Psychedelic Experience (SOCQ) | ~24 h after the dosing session
  States of Consciousness Questionnaire (SOCQ) selected domains (pre-specified) to characterize phenomenology beyond MEQ-30 and explore correlations with antidepressant outcomes.
Psychological Flexibility - AAQ-10 | Baseline to Week 4; Baseline to Week 6
  Change in Acceptance and Action Questionnaire (10- item) score from baseline to Week 4 and Week 6; exploratory correlations with ΔMADRS and 5D-ASC/SOCQ.
Altered States of Consciousness Phenomenology (5D-ASC) | 24 hours after the dosing session
  Change in 5-Dimensions Altered States of Consciousness (5D-ASC) total and domain scores to assess the global and detailed phenomenology of the psychedelic experience and to explore correlations with antidepressant outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Francisney P Nascimento, 1, Study Director — Federal University of Latin American Integration
Locations (1):
- Federal University of Latin American Integration, Foz do Iguaçu, Paraná, Brazil